CLINICAL TRIAL: NCT04634487
Title: Polish Registry of Takotsubo Syndrome
Acronym: Pol-Tako
Status: Recruiting | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Monika Budnik, Principal Investigator, Medical University of Warsaw
Other Study IDs: Pol-Tako
Record Dates: First submitted 2020-10-09; First posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Takotsubo Syndrome
MeSH Terms: conditions — Takotsubo Cardiomyopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Polish registry of takotsubo syndrome

ELIGIBILITY:
Inclusion Criteria:

all patients with takotsubo syndrome

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalised with takotsubo syndrome in Poland
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with in-hospital complications and mortality | through study completion, an average of 1 year
  In hospital complications include atrial fibrillation, ventricular tachycardia, ventricular fibrillation, atrioventricular block, cardiogenic shock, cardiac arrest

SECONDARY OUTCOMES:
Number of participants with complications with echocardiography | through study completion, an average of 1 year
  Complications include: severe mitral regurgitation, fluid in the pericardium, right ventricle disfunction, ventricular septum rupture

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided